CLINICAL TRIAL: NCT02484612
Title: Effect of Acute Exercise Intensity on Energy Intake in Adolescents: Effect of Weight Status
Brief Title: Exercise Intensity and Appetite in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Blaise Pascal, Clermont-Ferrand (Other)
Responsible Party: Principal Investigator, THIVEL David, PhD, As/Pr, Research scientist, Université Blaise Pascal, Clermont-Ferrand
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: AME2P Laboratory
Record Dates: First submitted 2015-06-19; First posted 2015-06-29 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean adolescents (Experimental): 15 lean adolescents (BMI Under the national cut-offs for obesity), 12-15 years old, males, will be recruited
  Interventions: Behavioral: acute exercise
- Obese adolescents (Experimental): 15 obese adolescents (BMI above the national cut-offs for obesity), 12-15 years old, males, will be recruited
  Interventions: Behavioral: acute exercise

INTERVENTIONS:
Behavioral: acute exercise

SUMMARY:
Acute exercise has been shown to affect subsequent energy intake in obese adolescents. Indeed, it has been shown several times that an intensive bout of exercise (above 70% of the individual maximal capacities) can reduce energy intake at the following meal in obese adolescents, with no modification of his appetite feelings.

Although this results has been replicated several times, it remains unknown if those nutritional adaptations are due to post-exercise modifications of some gastro-peptides implicated in appetite control, as detailed in adults.

The aim of this work is to question whether or not post-exercise energy intake is explained by appetite-regulating hormones that are affected by the exercise bout in both lean and obese youth.

DETAILED DESCRIPTION:
After an first medical visit to ensure that the adolescents have the ability to complete the whole study, the participants will have to complete several clinical examinations:

* anthropometric measurements
* Body composition assessed by dual energy x-ray absorptiometry
* Maximal aerobic test

They will then randomly complete the following conditions:

* CON: a control day without exercise;
* HIE: an exercise day with an exercise set at 75% of the capacities
* LIE: an exercise day with an exercise set at 40% of the capacities

The exercises or the rest condition will be done by the end of the morning and a buffet meal will be proposed during which the participants will be asked to eat as much as wanted.

Blood samples will be drawn before, after, 15 after and 30 minutes after the exercise to assess the main appetite regulating hormones involved in appetite regulation (PYY, Cholecystokinin ...) appetite feelings will be assessed throughout the day at regular interval using visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 15 years old adolescents
* Obese according to international values for BMI
* Being registered to the national social security insurance
* no eating disorders
* no medications
* metabolic disorders

Exclusion Criteria:

* metabolic disorders
* food disorders
* physical disability

Ages: 12 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
energy intake in kcal | up to 2 months
  buffet meal